CLINICAL TRIAL: NCT05439759
Title: Characterization of Multiple Factors in Training and Plasticity in Central Vision Loss: Healthy Vision
Brief Title: Factors in Learning And Plasticity: Healthy Vision
Acronym: FLAP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of California, Riverside (Other)
Responsible Party: Principal Investigator, Kristina M Visscher, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 300006197 (Study 1)
Record Dates: First submitted 2022-06-07; First posted 2022-06-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Central Visual Impairment; Macular Degeneration
Keywords: plasticity; central vision loss; perceptual learning
MeSH Terms: conditions — Blindness, Cortical; Macular Degeneration; Scotoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Condition 1: Training visual sensitivity (Experimental): A standard Perceptual Learning approach to train early visual processes of discriminating the orientation of Gabor patches presented at threshold- level contrast. Preliminary data, using this method, in normally seeing and MD participants show both feasibility and preliminary evidence that this training gives rise to improvements in acuity.
  Interventions: Behavioral: Condition 1: Training visual sensitivity
- Condition 2: Training spatial integration (Experimental): Most visual tasks involve integrating features to discriminate objects, therefore requiring brain areas that can integrate features from multiple receptive fields from early visual areas. Thus spatial integration involves what investigators refer to as mid-level vision. Spatial integration is a particular concern in developing a PRL since an area of the visual periphery that is best suited to discriminate a simple visual feature may not be appropriate to integrate information across objects, such as in reading or recognizing facial identity or expression. Investigators address this issue with a targeted spatial integration training approach developed by MPI Seitz and based on contour integration tasks used in previous PL studies to train mid-level visual processes. Target stimuli consist of contours formed by spaced Gabors. Difficulty of detecting the target is manipulated by varying orientation jitter of Gabors making up the target.
  Interventions: Behavioral: Condition 2: Training spatial integration
- Condition 3: Training spatial attention (Experimental): A key attribute of most real-world visual tasks is that individuals alternate shifting and holding attention and eye movements to different objects in the visual field while searching for and discriminating possible sources of visual information. To train this, investigators will implement a task structure that requires participants to alternate between holding and switching attention and making targeted eye movements. The basic task is to press a key whenever a red circle appears in a series of other colored circles, with a target presented every 2 to 4s. Participants must maintain vigilance for relatively long periods, detect objects in the near periphery, switch attention based upon exogenous and endogenous cues, and make eye- movements to move areas of spared vision to those locations. These are aspects of attention and eye movements not incorporated in Conditions 1 and 2.
  Interventions: Behavioral: Condition 3: Training spatial attention
- Condition 4: Combination training (Experimental): In Condition 4, investigators combine the elements of Conditions 1-3. The investigators test the extent to which a combined training gives rise to the joint benefits of each training individually, or integrative benefits potentially surpass the benefits of the individual training alone. The visual sensitivity task from Condition 1 will alternate across blocks with the spatial integration task from Condition 2, using the timing of targets and location switches from Condition 3; Gabors or contours are used as targets instead of the red- circle in Condition 3 and a fixation point is presented instead of distractors to maintain a similar stimulus configuration as Conditions 1 and 2.
  Interventions: Behavioral: Condition 4: Combination training

INTERVENTIONS:
Behavioral: Condition 1: Training visual sensitivity — Investigators adopt a standard PL approach to train early visual processes of discriminating the orientation of Gabor patches presented at threshold contrast. Across training blocks, Gabors will range in spatial frequency, where contrast is adapted with a 3/1 staircase. Whenever a specific contrast threshold is reached, spatial frequency will increase by 2 cycles per degree and contrast will be reset. Preliminary data from this method in normally seeing and MD participants show both feasibility and tentative evidence that this training gives rise to improvements in acuity.
  Arms: Condition 1: Training visual sensitivity
Behavioral: Condition 2: Training spatial integration — Spatial integration involves what the investigators refer to as mid-level vision. Spatial integration is a concern in developing a PRL since an area of the visual periphery that is best suited to discriminate a simple visual feature may not be appropriate to integrate information across objects, such as in reading or recognizing facial identity or expression. The investigators address this issue with a targeted spatial integration training approach developed by MPI Seitz and based on contour integration tasks used in previous PL studies to train mid-level visual processes. Target stimuli consist of contours formed by spaced Gabors. The difficulty is manipulated by varying orientation jitter of Gabors. Several optotypes will be included to promote generalization, including shapes and facial expressions.
  Arms: Condition 2: Training spatial integration
Behavioral: Condition 3: Training spatial attention — The investigators will implement a task structure that requires participants to alternate between holding and switching attention and making targeted eye movements. The basic task is to press a key whenever a red-circle appears in a series of other colored-circles, with a target presented every 2 to 4s. Participants must maintain vigilance for relatively long periods, detect objects in the near periphery, switch attention based upon exogenous and endogenous cues, and make eye- movements to move areas of spared vision to those locations. These are aspects of attention and eye movements not incorporated in Conditions 1 and 2.
  Arms: Condition 3: Training spatial attention
Behavioral: Condition 4: Combination training — Daily tasks involve a combination of being sensitive to basic visual features, being able to integrate these features, and directing attention and eye movements to better evaluate the information of potential interest. To address this integrative nature of real-world vision,Condition 4 combines the elements of Conditions 1-3.
  Arms: Condition 4: Combination training

SUMMARY:
A greater understanding of plasticity after central vision loss can inform new therapies for treating low vision and has the potential to benefit millions of individuals suffering from low vision. The treatment of low vision is particularly relevant to the mission of the National Eye Institute (NEI) to support research on visual disorders, mechanisms of visual function, and preservation of sight. The comparison of different training and outcome factors is in line with the National Institute of Mental Health (NIMH) Research Domain Criteria (RDOC) framework and studies in an aging population are consistent with the mission of the National Institute on Aging (NIA).

DETAILED DESCRIPTION:
Research on perceptual learning (PL) has been dominated by studies that seek to isolate and improve individual visual processes. However, an important translational outcome of PL research is to address the needs of patients with vision loss, who seek to improve performance on daily tasks such as reading, navigation, and face recognition. These more ecological cases of behavioral change and cortical plasticity, which are inherently complex and integrative, have revealed significant gaps in a more holistic understanding of how multiple visual processes and their associated brain systems jointly contribute to durable and generalizable PL. To address these gaps, here the investigators study simulated and natural central vision loss. The investigators focus on macular degeneration (MD), one of the most common causes of vision loss (projected to affect 248 million people worldwide by 2040), which results from damage to photoreceptors in the macula that disrupts central vision. Such central vision loss is a superb lens through which study to how ecologically relevant changes in the use of vision relate to changing brain activity and connectivity because it represents a massive alteration in visual experience requiring reliance on peripheral vision for daily tasks. With the use of eye-trackers and gaze-contingent displays that induce central scotomas, central vision loss can be simulated in normally seeing individuals, who then develop peripheral looking patterns that resemble compensatory vision strategies seen in MD patients. Ideal use of peripheral vision requires improvement in multiple vision domains, three of the most important being: early visual processing (e.g., visual sensitivity), mid-level visual processing (e.g., spatial integration), and attention and eye-movements. To date, no study has systematically investigated these three domains of PL and their neural underpinnings. The proposed research plan rests on rigorous prior work showing that PL influences multiple brain structures and functions related to these three domains. The investigators propose a novel approach of systematically measuring how different training regimes related to the three domains influence a broad range of psychophysical and ecological behaviors (Aim 1), how these changes arise from plasticity in brain structure and function (Aim 2), and how PL after simulated central vision loss compares to PL in MD (Aim 3). This work is significant and innovative as it will be the first integrated study of PL characterizing multiple trainable factors and their impact on diverse behavioral outcomes and on cutting-edge assessments of neural representations and dynamics. It is also the first study to directly compare PL in MD patients with PL in a controlled model system of central visual field loss with simulated scotomas, which if validated will allow the use of this model system to interrogate MD in larger samples of healthy individuals. The Investigators will also share a unique dataset that will help the field to understand behavioral and neural plasticity after central vision loss and individual differences in responsiveness to training. Finally, this work will illuminate basic mechanisms of brain plasticity after sensory loss that may generalize to other forms of rehabilitation after peripheral or central damage.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30
* Corrected vision (20/40 or better)
* No reported incidence of retinal pathology.

Exclusion Criteria:

* Pacemaker or any ferromagnetic metal implanted in their body
* Metal of any type implanted in their head (limited dental work is acceptable)
* Claustrophobia
* Needing non-standard glasses (other than the simple MR-compatible glasses that can be supplied) for best-corrected distance vision
* Being hearing-impaired
* Weight over 300 pounds
* Maximum body girth over 60 inches
* Previous serious head injury
* Presence of hallucinations or delusions
* Excessive old, or colorful tattoos, especially near the head
* Pregnancy
* Braces/permanent retainer

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Radial Bias from the Crowding Task after completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  The ratio of the crowding threshold along the axis connected to the fovea vs. along the orthogonal axis.
Change from Baseline Saccadic Precision after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Consistency across trials in placement of the first saccade calculated by the distribution across trials (bivariate contour ellipse area) of the landing point of the first fixation of each trial.
Change from Baseline Fixation Stability after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Normalizing fixations in the PRL to the first fixation to that region and calculating the distribution of all fixation locations in this normalized space (measured as a bivariate contour ellipse area).

OTHER OUTCOMES:
Change from Baseline Acuity after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Acuity threshold from the Landolt C task.
Change from Baseline Contrast Sensitivity after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Threshold value from contrast sensitivity task.
Change from Baseline Minimal print size from the MNREAD task after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Minimal print size from the MNREAD task
Change from Baseline Precision of Reconstructed Representation of Stimulus Orientation after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Precision of reconstructed representation of stimulus orientation (quantified with FWHM)
Change from Baseline Population receptive field size in V1, V2 and V3 representations of URL and PRL after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Population receptive field size in V1, V2 and V3 representations of URL and PRL (quantified as PRF sigma in the swath of cortex associated with that retinal location).
Change from Baseline Cortical thickness in V1, V2 and V3 representations of the PRL and URL after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Cortical thickness in V1, V2 and V3 representations of the PRL and URL (quantified as mm of cortical thickness)
Change from Baseline Orientation jitter threshold in the contour integration task at PRL or URL after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Orientation jitter threshold in the contour integration task (quantified as threshold average jitter) at PRL or URL.
Change from Baseline Crowding Threshold after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  In the contour integration task stimuli are untrained contours of alphanumeric characters made of Gabor elements. This test allows us to estimate how the magnitude of crowding may change at the PRL compared to the non-PRL.
Change from Baseline Decoding classification accuracy for an attended character after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Decoding classification accuracy for an attended character, based on decoding from MRI data within VWFA and LOC regions of interest.
Change from Baseline Strength of background connectivity between areas with larger receptive fields (V4) to the smaller receptive fields contributing information to that area. after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  This is measured as functional connectivity (z-transformed Pearson's r) between voxels in V1 to voxels in V4 in that represent the same portion of retinotopically mapped space. Measured in portions of cortex representing PRL and URL.
Change from Baseline Sustained Attention after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Reaction time of detection of orientation of Landolt Cs presented in an RSVP stream at the beginning of each trial.
Change from Baseline Endogenous Attention after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Endogenous attention: reaction time when switching between locations due to an endogenous cue on valid vs nonvalid trials.
Change from Baseline Exogenous Attention after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Exogenous attention: reaction time when switching between locations due to an exogenous cue on valid vs. nonvalid trials.
Change from Baseline Saccadic Re-referencing after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Saccadic Re-referencing: number of first fixations that do not cover the target location with the scotoma.
Change from Baseline Decoding classification accuracy for decoding the locus of spatial attention (PRL or URL), regardless of stimulus type after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Decoding classification accuracy for decoding the locus of spatial attention (PRL or URL), regardless of stimulus type. This will be examined in frontal (FEF), parietal (SPL/IPS) and higher order visual (LOC) regions.
Change from Baseline Top-down modulation of visual areas after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Top-down modulation of visual areas: background connectivity between frontoparietal control regions (FEF, SPL/IPS) and visual areas ( V1, V2, V3).
Change from Baseline Reading speed in the MNREAD task after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Reading speed in the MNREAD task (words per minute).
Change from Baseline Completion time in the trail making task after Completion of Training at approximately 7 weeks | Baseline and Within 3 weeks of training completion, training is complete 7 weeks from baseline on average
  Completion time in the trail making task

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UAB, Birmingham, Alabama
  - University of California, Riverside, Riverside, California

IPD SHARING:
Plan to Share IPD: Yes
Plan Description: Results of the project will be submitted to the relevant repository (ClinicalTrials.gov, or Open-ScienceFramework, MRI data to OpenfMRI) within one year of the final participant completing data collection. The investigators expect to report participant flow by group (intervention or control), participant demographics (age, sex assigned at birth, years of education), outcome measures and statistical analyses, adverse events (if applicable), and limitations or caveats of our results. The investigators also will ensure that the final protocol and statistical analysis code are uploaded to the record. No Protected Health Information will be shared.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Within one year of the final participant completing data collection.